CLINICAL TRIAL: NCT03064906
Title: Evaluating Meal Performance and Effect of Moderate Intensity Exercise in Patients With Type 1 Diabetes With the Insulet Automated Glucose Control System: IDE 2
Brief Title: Insulet Artificial Pancreas Evaluating Meal Performance and Moderate Exercise (IDE2)
Acronym: IDE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IDE2
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D, Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The two-part study schedule consists of a 7±1 day outpatient, open-loop phase, followed by one 54-hour (Option A - Meal Performance and/or Option B - Exercise), hybrid closed-loop phases conducted in a supervised CRC or hotel/rental house setting. Subjects may participate in hybrid closed-loop session Option A and/or Option B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Meal Performance and/or Exercise (Other): This study is a two-part, multi-center, observational clinical trial being conducted in a Clinical Research Center (CRC) setting using the Insulet AP (artificial pancreas) system.
  Subjects may participate in hybrid closed-loop session Option A - Meal Performance and/or Option B - Exercise, but are not required to participate in both. If participating in both, Option A and Option B must be conducted in separate sessions.
  Interventions: Device: Insulet AP (artificial pancreas) System

INTERVENTIONS:
Device: Insulet AP (artificial pancreas) System — Insulet AP (artificial pancreas) system, using the Omnipod® insulin management system, Dexcom G4 Share® AP System and personalized model predictive control algorithm.

SUMMARY:
To assess the safety and performance of the Insulet AP (artificial pancreas) system, using the Omnipod® insulin management system, Dexcom G4 Share® AP System and personalized model predictive control algorithm in adults with type 1 diabetes consuming high fat meals and undertaking moderate intensity exercise.

DETAILED DESCRIPTION:
The two-part study schedule consists of a 7±1 day outpatient, open-loop phase, followed by one 54-hour, hybrid closed-loop phases conducted in a supervised CRC or hotel/rental house setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 18.0 to 65.0 years
2. Diagnosed with type 1 diabetes for at least one year. Diagnosis is based on investigator's clinical judgment.
3. Total daily dose (TDD) of insulin ≥0.3 units/kg/day and A1C >6% at screening
4. Currently using an insulin pump with U-100 rapid-acting insulin analogs and on pump therapy for at least 6 months prior to study start
5. Willing to use the study CGM device for the duration of the study
6. Willing to use the Omnipod® Insulin Management System during the study
7. Willing to perform all fingerstick BG testing with the study-approved glucose meter at the frequency specified in the study protocol
8. Willing to abide by meal recommendations for breakfast, lunch and dinner during the study
9. Willing to participate in moderate intensity exercise for up to 45 minutes if taking part in Option B
10. Willing to refrain from use of acetaminophen and supplemental vitamin C (>2000 mg/daily) for the entire duration of participation in the study
11. Willing and able to sign the Informed Consent Form (ICF)

Exclusion Criteria:

1. A1C >10% at the screening visit
2. One or more episodes of severe hypoglycemia requiring emergency room (ER) visit or hospitalization within the past 6 months
3. Hypoglycemic unawareness as determined by a score of ≥4 "R" responses on the Clarke Questionnaire
4. One or more episodes of diabetic ketoacidosis requiring ER visit or hospitalization within the past 6 months
5. Used non-insulin anti-diabetic medication within last 30 days
6. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD or implant)
7. Dermatological conditions at the proposed sensor wear sites that in the investigator's opinion could preclude ability to wear the Pod and/or the Dexcom sensor
8. Current or known history of cardiovascular disease, arrhythmia, myocardial infarction (MI) or stroke. An electrocardiogram (ECG) must be obtained within 6 months.
9. Currently undergoing systemic treatment with steroids or immunosuppressive medication
10. Current illness that would interfere with participation in the study
11. Currently participating in another clinical study using an investigational drug or device
12. Recent (within the preceding 30 days) participation in a clinical study using an investigational drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Percentage of time in hypoglycemic range (defined as < 70 mg/dL) | 54 hours
Percentage of time in hyperglycemic range(defined as ≥ 250 mg/dL) | 54 hours

SECONDARY OUTCOMES:
Mean glucose | 54 hours
Percentage of time < 50 mg/dL | 54 hours
Percentage of time < 60 mg/dL | 54 hours
Percentage of time > 180 mg/dL | 54 hours
Percentage of time ≥ 300 mg/dL | 54 hours
Percentage of time between 70-180 mg/dL | 54 hours
Percentage of time between 70-140 mg/dL | 54 hours
Standard deviation | 54 hours
Coefficient of variation | 54 hours
Meal challenge-12 hour PPG dinner | 54 hours
  The post-prandial glucose response including time to peak glucose, peak glucose concentration, and peak glucose excursion and the 12-hour post-prandial period following dinner.
Meal challenge-4 hour PPG breakfast | 54 hours
  The post-prandial glucose response including time to peak glucose, peak glucose concentration, and peak glucose excursion for the 4-hour post-prandial period following breakfast.
Meal challenge-4 hour PPG lunch | 54 hour
  The post-prandial glucose response including time to peak glucose, peak glucose concentration, and peak glucose excursion for the 4-hour post-prandial period following lunch.
Exercise challenge-immediate and delayed glucose response | 54 hour
  The immediate (2 hours) and delayed (24 hours) glucose response to moderate intensity exercise.
Effect of changing setpoints | 54 hour
  Effect of changing setpoints to overall performance.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Diablo Clinical Research, Walnut Creek, California
  - University of Colorado Denver, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No